CLINICAL TRIAL: NCT03020511
Title: Effects of Ancient Grains-based Diet in a Closed Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACPM19
Record Dates: First submitted 2016-12-30; First posted 2017-01-13 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Gluten Sensitivity
Keywords: Modern grains; ancient grains; immunologic response; microbiota
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ancient wheat flours (Other): We prospectively will survey 30 nuns from the "Congregazione delle Suore Collegine della Santa Famiglia", Palermo, Italy. The subjects will be recruited between January 2017 and June 2017 and will be examined before and after the diet period (30 days) with ancient grains, undergoing clinical evaluation and blood and feces samples collection. Ancient wheat flours will be administered in open label for 30 days
  Interventions: Other: Ancient wheat flours

INTERVENTIONS:
Other: Ancient wheat flours — Ancient wheat flours will be administered in open label for 30 days

SUMMARY:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. It is also believed that this condition is worldwide increasing, due to the evolution of wheat breeding (i.e. consumption of wheats with high gluten content), and that "ancient" wheat flour varieties are better tolerated by NCWS patients than the "modern" ones. This effect could be related to a lower immunogenic stimulation of the ancient wheat than the modern ones. The aim of the study is to evaluate the effect of a diet based on ancient grains in a "closed" community (i.e. nuns from enclosed religious order) as regard to 1) main haematochemical parameters and vitamins, 2) intestinal microbiota (bacterial flora), and 3) cytokines production from peripheral blood mononuclear cells (PBMC), before and after the diet period (30 days) with ancient grains.

DETAILED DESCRIPTION:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. Therefore, NCWS pathogenesis has been attributed to very different mechanisms: innate or adaptive immunity, non IgE-mediated food allergy, amylase/trypsine inhibitors pro-inflammatory effects, incomplete digestion and/or absorption of fermentable oligosaccharides and disaccharides, monosaccharides and polyols, and, finally, psychological effect. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). It is also believed that this condition is worldwide increasing, due to the evolution of wheat breeding (i.e. consumption of wheats with high gluten content), and that "ancient" wheat flour varieties are better tolerated by NCWS patients than the "modern" ones. More in details, it has been demonstrated that in patients with NCWS foods containing modern (i.e. "Manitoba") wheat flour varieties may trigger immunological mechanisms of inflammation (i.e. CXCL10 secretion) and may alter intestinal permeability; on the contrary, these effects was not observed with wheat flour from ancient (i.e. "Kamut" or "Senatore Cappelli") varieties. Therefore, the aim of the study is to evaluate the effect of a diet based on ancient grains (i.e. a mixture of "Tumminia", "Perciasacchi", "Senatore-Cappelli" and "Margherito" grains) in a "closed" community (i.e. nuns from enclosed religious order) as regard to: 1) main haematochemical parameters and vitamins (serum creatinine, serum glutamic-oxaloacetic transaminase, serum glutamic-pyruvic transaminase, hemoglobin, serum iron, serum ferritin, blood glucose, serum sodium, total cholesterol, glycated hemoglobin, vitamin B12, and vitamin D), 2) intestinal microbiota (bacterial flora), and 3) cytokines production from peripheral blood mononuclear cells (PBMC), before and after the diet period (30 days) with ancient grains.

ELIGIBILITY:
Inclusion Criteria:

* Nuns from the "Congregazione delle Suore Collegine della Santa Famiglia", Palermo, Italy.

Exclusion Criteria:

* N/A

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Laboratory Values evaluation | Change from baseline at 30 days
  Laboratory Values evaluation at baseline and after a 30 days challenge with ancient grains-based diet.

SECONDARY OUTCOMES:
Intestinal microbiota (bacterial flora) by feces samples examination | Change from baseline at 30 days
  Evaluation of modifications of intestinal microbiota (bacterial flora) by feces samples examination, before and after a 30 days challenge with ancient grains-based diet.
Cytokines production from PBMC | Cytokines production from PBMC after the diet period (30 days) with ancient grains
  Evaluation of modifications in cytokines production from PBMC, before and after the diet period (30 days) with ancient grains.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (1):
- Congregazione delle Suore Collegine della Santa Famiglia, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Valerii MC, Ricci C, Spisni E, Di Silvestro R, De Fazio L, Cavazza E, Lanzini A, Campieri M, Dalpiaz A, Pavan B, Volta U, Dinelli G. Responses of peripheral blood mononucleated cells from non-celiac gluten sensitive patients to various cereal sources. Food Chem. 2015 Jun 1;176:167-74. doi: 10.1016/j.foodchem.2014.12.061. Epub 2014 Dec 23. PMID 25624220